CLINICAL TRIAL: NCT00152750
Title: Aggressive Behaviour in Children With Tourette's Syndrome (TS) and Comorbid Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Study of Clonidine on Sleep Architecture in Children With Tourette's Syndrome (TS) and Comorbid ADHD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: StephensClonidine2005; SickKids #XG05-032; REB 130/2004
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2006-10

CONDITIONS: Tourette's Syndrome; Attention Deficit Hyperactivity Disorder
Keywords: Tourette's Syndrome; Attention Deficit Hyperactivity Disorder; Children; Sleep disorders; Aggression
MeSH Terms: conditions — Tourette Syndrome; Attention Deficit Disorder with Hyperactivity; Sleep Wake Disorders; Aggression

INTERVENTIONS:
Drug: APO-clonidine

SUMMARY:
In the present study, we examine the question "Will day-time aggression in children improve when their night-time sleep is treated with pharmacological intervention (i.e. clonidine)?" There is considerable anecdotal evidence that clonidine may provide an effective alternative to neuroleptics for treating aggression in children -- first by improving the overall quality of their sleep, and second by providing a safer and more readily tolerated medication with fewer side-effects and a greater probability of long-term compliance. This study uses a double blind placebo controlled design to gather scientific evidence that will help elucidate the mechanisms underlying this treatment effect and will help clarify the relationship between sleep disorders and aggression in children. Our results are expected to help physicians make informed treatment decisions regarding the use of clonidine to improve the quality of sleep and possibly treat problems with aggression in their pediatric patients

DETAILED DESCRIPTION:
Background: Childhood sleep disturbance is pervasive, yet remains under-treated and one of the most poorly researched areas in pediatric psychopharmacology. Of particular concern is the growing evidence of an association between sleep disturbance and aggression in children. Childhood aggression is a serious public health problem and predicts adolescent delinquency, academic difficulties and truancy, and substance abuse. Children with Tourette's syndrome (TS) and co-morbid attention deficit hyperactivity disorder (ADHD) will be studied in a trial of a common pharmacological treatment (clonidine) that is expected to improve sleep architecture and thereby clarify the relation between sleep disturbance and aggression.

Hypothesis: Our main hypothesis is that improvement in children's sleep will be associated with a reduction in their aggression and an increase in their daily function.

Method: A double-blind placebo controlled trial with 32 subjects (aged 9-14 years) with diagnoses of TS & co-morbid ADHD. Subjects will undergo a mental health assessment, ECG, laboratory testing and 2-night polysomnography (sleep study) at baseline. Subjects will then be randomized to a treatment (clonidine) or placebo group for an 8-week trial. Clonidine will be titrated and subjects monitored weekly. A second 2-night sleep study and mental health assessment will occur at trial end.

Expected results: We expect an improvement in the initial onset, duration and overall sleep quality in the treatment group (clonidine), with a resulting decrease in daytime aggression and increase in daily overall level of functioning; sleep and aggression in the placebo group are not expected to improve.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* Meet the DSM-III-R criteria for Tourette syndrome based on the assessment of a study psychiatrist and the presence of comorbid Attention Deficit Hyperactivity Disorder (ADHD) according to DSM-IV diagnostic criteria
* A negative history of psychiatric illness that requires treatment.
* Medication free for a minimum period of six (6) weeks at the time of entry into the study
* Between the ages of 9:0 years and 14:11 years
* An initial screening score on the Children's Aggression Scale-Parents Version of at least +1SD above average on at one or more of the four subscales.
* Adequate English language comprehension and production (sufficient to respond to questions from the investigators)
* Be able and willing to cooperate with the study protocol
* All parents/caregivers will provide consent and subjects (children/adolescents) will give their informed assent prior to participating in any study procedures.
* Known history of sleep disturbances (children will be considered to experience sleep disturbances if their sleep latency regularly exceeds 30 minutes; to have a general poor quality of sleep if there are frequent awakenings (>2 nightly), nightmares or restlessness; or if they experience difficulty awakening, marked difficulty with arousal or consistent oversleeping. For the purposes of this study, a disturbance in sleep is considered only if it is chronic (lasting more than one month) and frequent (two or more times per week).

Exclusion Criteria:

*Evidence of Pervasive Developmental Disorder, known seizure disorder, history of severe head trauma, post-traumatic stress disorder, depression, known organic basis for a sleep disorder and/or an estimated Full Scale Intellectual Quotient below 85

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32
Dates: Start 2006-09; Study Completion 2008-10

PRIMARY OUTCOMES:
Objective: The differences between baseline and final polysomnographic sleep architecture measurements.

SECONDARY OUTCOMES:
Subjective:Differences in scores from baseline to trial end on the Sleep Disturbance Scale for Children, the Children's Sleep habits Questionnaire, and scales of Aggressive or maladaptive behaviour (Parent,Teacher and Self reports).

CONTACTS AND LOCATIONS:
Overall Officials: Robyn J Stephens, PhD.C.Psych., Principal Investigator — Youthdale Treatment Centres
Locations (1):
- Youthdale Treatment Centres, Toronto, Ontario, Canada

REFERENCES:
- See also: Youthdale Treatment Centres — http://www.youthdale.ca